CLINICAL TRIAL: NCT06209112
Title: Feasibility and Safety of an Over-pressure wash-in Method Using Fresh Gas Flow 0.5 L and Sevoflurane 8% During Initiation of Low-flow Anaesthesia: a Prospective, Randomised, Description Study
Brief Title: Sevoflurane Wash in Method Using Conventional Flows Versus Low Flows of 0.5L
Status: Completed | Type: Observational
Sponsor: Royal Hospital, Oman (Other Government)
Responsible Party: Principal Investigator, Harihar V Hegde, Consultant, Department of Anesthesia & Intensive Care, The Royal Hospital, Royal Hospital, Oman
Other Study IDs: MoH/CSR/23/27624
Record Dates: First submitted 2024-01-06; First posted 2024-01-17 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Inhalation; Gas
MeSH Terms: conditions — Respiratory Aspiration; Mucopolysaccharidosis IV | interventions — Sevoflurane

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Conventional group' (Group C): The 'conventional' group (Group C): FGF will be set to 6 L/min and the FVS 3% at Tzero. The FGF will be reduced to 0.5 L/min upon reaching FAS 2%. Hereafter, the FVS will be set to 4% and maintained till 15 min (T15) from Tzero.
  Interventions: Drug: Sevoflurane
- Over-pressure group' (Group OP): The 'over-pressure' group (Group OP): FGF will be set to 0.5 L/min and FVS 8% at Tzero.
  Subsequently, the FVS will be set to 4% upon reaching FAS 2% and maintained till 15 min (T15) from Tzero.
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Sevoflurane — The time of reaching FAS=2% will be noted in both the groups. The time taken in seconds from Tzero to reach FAS 2% (Ttarget) will be calculated. Inspired concentration of Sevoflurane (FIS), FAS, and age-adjusted MAC will be retrieved from the automatically recorded 'trend' of parameters. FIS, FAS and age-adjusted MAC will be noted every 30 sec. starting from Tzero, till T5 and every minute thereafter until T15.

SUMMARY:
The goal of this observational study is to to evaluate a technique of initiating Sevoflurane low-flow anesthesia which is simple, has a quick wash-in and minimises gas consumption without compromising the safety when compared to conventional method of attaining low-flow anesthesia using initial high flows.

Participants will explained about the procedure of induction of general anesthesia using either one of the above two methods and written consent will be obtained prior to inclusion in the study.

DETAILED DESCRIPTION:
After obtaining the approval from the Institutional Ethics Committee of The Royal Hospital, Muscat, we will register this prospective, randomised, descriptive study in an appropriate online clinical trial registry. A written informed consent will be obtained from all the patients. Forty-eight patients of either gender aged 18-65 years, with American Society of Anesthesiologists (ASA) physical status of 1-2, undergoing elective surgery with the expected duration more than 1 hour under general anaesthesia requiring endotracheal intubation will be included. Pregnant women, smokers, patients with a body mass index (BMI) ≥30 kg/m2, cardiac/pulmonary/renal or liver impairments, upper or lower respiratory infections within the past 6 weeks and anticipated difficult airway will be excluded.

Age, gender, height and weight of the patients will be recorded. All the patients will follow the standard fasting requirements and receive no sedative premedication. They will be randomised before entering the operating room into one of the two groups, 'conventional group' (Group C) and 'over-pressure group' (Group OP), using block randomisation technique with varying block sizes. An appropriate intravenous cannula will be secured in the operating room and Ringer's Lactate 500 ml will be started. The patients will receive standard anaesthetic care and intra-operative monitoring with electrocardiogram, pulse oximeter (SpO2), non-invasive blood pressure (NIBP) and capnography. Anaesthesia workstation (GE Healthcare, Madison, WI, USA) which has an integrated anaesthetic gas analyser, displays age-adjusted MAC according to the internal algorithm and returns sampled gas to the breathing system will be used in this study. The breathing system will consist of a 2 litres reservoir bag, disposable breathing circuit, heat-moisture exchanger and standard circle system with Sodalime as the CO2 absorbent. The workstation will be tested to ensure no leak in the system and vapourisers are calibrated.

Ideal Body Weight (IBW) of the patient will be calculated based on the following formula: IBW (kg)=50 + 0.91 (height in cm - 152.4) for Men and 45.5 + 0.91 (height in cm - 152.4) for Women. The ventilator will be preset in Pressure Control-Volume Guarantee (PCV-VG) mode with a tidal volume of 8 ml/kg of IBW, respiratory rate=14 breaths/min, positive end-expiratory pressure (PEEP)=5 cmH2O and an inspiratory:expiratory ratio of 1:2. The set minute volume will be noted. The alarm for end-tidal Sevoflurane (FES) will be set at 2% to alert the clinician.

Heart rate (HR), blood pressure (BP) and peripheral oxygen saturation will be recorded before induction of anaesthesia, every minute until 5 min after induction and every 5 min intervals thereafter. The FGF will be set at 6 L/min with 100% O2 during pre-oxygenation and manual ventilation. Following pre-oxygenation for 3 min, general anaesthesia will be induced with intravenous Fentanyl 2 μg/kg followed by Propofol 2 mg/kg administered over 30 seconds and Rocuronium 1 mg/kg for neuromuscular blockade. Lungs will be ventilated manually and propofol 20 mg every minute will be administered until tracheal intubation. Tracheal intubation with an appropriate size endotracheal tube (ETT) will be performed 90 seconds later, the cuff inflated to 25-30 cmH2O using a cuff-pressure monitor device and ETT secured with an adhesive tape. The correct ETT position will be confirmed by auscultation and square-wave capnography. FGF will be paused during intubation and restarted after inflating the ETT cuff. The FGF hereafter will consist of O2 and Air with a set FIO2=0.6. FGF and Sevoflurane vapouriser dial (FVS) will be set as per the group allocation and mechanical ventilation will begin. The time of opening of vapouriser will be considered Tzero.

Following will be the steps during wash-in for achieving LFA:

The 'conventional' group (Group C): FGF will be set to 6 L/min and the FVS 3% at Tzero. The FGFwill be reduced to 0.5 L/min upon reaching FAS 2%. Hereafter, the FVS will be set to 4% andmaintained till 15 min (T15) from Tzero.

The 'over-pressure' group (Group OP): FGF will be set to 0.5 L/min and FVS 8% at Tzero. Subsequently, the FVS will be set to 4% upon reaching FAS 2% and maintained till 15 min (T15) from Tzero.

The time of reaching FAS=2% will be noted in both the groups. The time taken in seconds from Tzero to reach FAS 2% target concentration (Ttarget) will be calculated. Inspired concentration of Sevoflurane (FIS), FAS, and age-adjusted MAC will be retrieved from the automatically recorded 'trend' of parameters. FIS, FAS and age-adjusted MAC will be noted every 30 sec. starting from Tzero, till T5 and every minute thereafter until T15.

Consumption of gases (Oxygen, Air and Sevoflurane) from the beginning until T15 will be retrieved. Any reduction in mean BP >20% from the baseline will be treated with intravenous Ephedrine 12 mg bolus and consumption of Ephedrine will be noted. Expired minute volume (MVE) at Ttarget and T15 will be noted. The study period will end at T15 in both the groups. Painting the surgical parts and draping will be permitted during the study period. Care will be taken to avoid any activity which risks ETT disconnection during the study period. Subsequent management of anaesthesia will be left to the discretion of the attending Anaesthesiologist.

For both the groups, 'stability of Sevoflurane concentration', defined as FAS in the target range of 1.6-2.4% during the time interval from Ttarget till T15 will be assessed. The investigator will be allowed during this period to increase or decrease if needed the vapouriser dial by 1% at a time every 2 min to keep the FES in the target range. The number of times the vapouriser dial is adjusted will be noted. The system will be considered 'stable' if the FAS is maintained in the target range without the need for dial adjustment and 'unstable' if vapouriser dial adjustment is needed at any time during this period. Delivery of Oxygen will be monitored to ensure at least 300 ml/min and delivered FIO2 at least 0.3 at all time. The investigator will be allowed to increase if needed the set FiO2 by 0.1 at a time every 2 min to keep the delivered FIO2>0.3. The number of times the set FIO2 is adjusted will be noted. End-tidal carbon dioxide (ETCO2) will be maintained <40.

For both the groups, 'stability of Sevoflurane concentration', defined as FAS in the target range of 1.6- 2.4% during the time interval from Ttarget till T15 will be assessed. The investigator will be allowed during this period to increase or decrease if needed the vapouriser dial by 1% at a time every 2 min to keep the FAS in the target range. The number of times the vapouriser dial is adjusted will be noted.

The system will be considered 'stable' if the FAS is maintained in the target range without the need for dial adjustment and 'unstable' if vapouriser dial adjustment is needed at any time during this period.

Delivery of Oxygen will be monitored to ensure at least 300 ml/min and delivered FIO2 at least 0.3 at all time. The investigator will be allowed to increase if needed the set FIO2 by 0.1 at a time every 2 min to keep the delivered FIO2>0.3. The number of times the set FIO2 is adjusted will be noted. Endtidal carbon dioxide (ETCO2) will be maintained between 30 and 40. The aim of the study is to assess during the wash-in phase of LFA the feasibility of the method, stability of the system and consumption of gases. The primary outcome will be the time required to achieve FAS 2%. Secondary outcomes will be the stability of the system assessed by the number of times vapouriser dial and the set FIO2 adjusted, consumption of gases and of ephedrine.

Statistical analysis Sample size is calculated based on a previous study8 which showed the 1-1-8 wash-in scheme with FGF=2L (O2 1 L + Air 1 L) and Sevoflurane dial at 8% yielded an FAS of 2% at 2 ± 0.5 min. Hence, we assume that with our wash-in technique using FGF=0.5 L (O2 + Air) and FVS 8% the time needed to reach FAS=2% will be around 8 min. To detect a difference of 2 min (25%) with standard deviation (SD) of 2 using an alpha level of 0.05 and a power of 0.90 the sample size needed is 22 per group. For a possible 10% dropouts, it is decided to include 24 patients per group.

Statistical analysis will be carried out using an appropriate statistical software. Data will be presented as mean ± SD or median (range). Intergroup differences will be assessed for significance using Student's t, Kruskal-Wallis, chi-squared or Fisher exact tests, as appropriate. P < 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status 1 and 2
* elective surgery with the expected duration more than 1 hour under general anaesthesia requiring endotracheal intubation

Exclusion Criteria:

* Pregnant women
* smokers
* patients with a body mass index (BMI) ≥30 kg/m2
* cardiac/pulmonary/renal or liver impairments
* upper or lower respiratory infections within the past 6 weeks and anticipated difficult airway will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Forty-eight patients of either gender aged 18-65 years, with American Society of Anesthesiologists (ASA) physical status of 1-2, undergoing elective surgery with the expected duration more than 1 hour under general anaesthesia requiring endotracheal intubation will be included.
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2024-01-30 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Time required to achieve alveolar concentration of sevoflurane at 2% | 15 minutes
  The primary outcome will be the time required to achieve FAS 2%.

SECONDARY OUTCOMES:
To know the stability of the circle system | 15 minutes
  Secondary outcomes will be the stability of the system assessed by the number of times vapouriser dial adjusted and number of times the set FIO2 adjusted, consumption of ephedrine and consumption of gases.

CONTACTS AND LOCATIONS:
Overall Officials: Harihar V Hegde, MD, Principal Investigator — The Royal Hospital, Oman
Locations (1):
- The Royal Hospital, Muscat, Muscat, Mucsat, Oman

IPD SHARING:
Plan to Share IPD: Undecided
Since the study group subjects are ASA physical status 1 and 2 patients, the patient data will not be valuable to any other researchers

REFERENCES:
- [Background] Baum JA. Low-flow anesthesia: theory, practice, technical preconditions, advantages, and foreign gas accumulation. J Anesth. 1999;13(3):166-74. doi: 10.1007/s005400050050. No abstract available. PMID 14530937
- [Background] Brattwall M, Warren-Stomberg M, Hesselvik F, Jakobsson J. Brief review: theory and practice of minimal fresh gas flow anesthesia. Can J Anaesth. 2012 Aug;59(8):785-97. doi: 10.1007/s12630-012-9736-2. Epub 2012 Jun 1. PMID 22653840
- [Background] Tribuddharat S, Sathitkarnmanee T, Vattanasiriporn N, Thananun M, Nonlhaopol D, Somdee W. 1-1-8 one-step sevoflurane wash-in scheme for low-flow anesthesia: simple, rapid, and predictable induction. BMC Anesthesiol. 2020 Jan 24;20(1):23. doi: 10.1186/s12871-020-0940-2. PMID 31980020
- [Background] Horwitz M, Jakobsson JG. Desflurane and sevoflurane use during low- and minimal-flow anesthesia at fixed vaporizer settings. Minerva Anestesiol. 2016 Feb;82(2):180-5. Epub 2015 Jul 22. PMID 26198766
- [Background] Jakobsson P, Lindgren M, Jakobsson JG. Wash-in and wash-out of sevoflurane in a test-lung model: A comparison between Aisys and FLOW-i. F1000Res. 2017 Mar 29;6:389. doi: 10.12688/f1000research.11255.2. eCollection 2017. PMID 28529707
- [Background] Upadya M, Saneesh PJ. Low-flow anaesthesia - underused mode towards "sustainable anaesthesia". Indian J Anaesth. 2018 Mar;62(3):166-172. doi: 10.4103/ija.IJA_413_17. PMID 29643549

DOCUMENTS (1):
  • Study Protocol (2023-12-26): https://cdn.clinicaltrials.gov/large-docs/12/NCT06209112/Prot_001.pdf